CLINICAL TRIAL: NCT04460781
Title: Post-Licensure Database Surveillance Study to Assess the Safety of Flublok Quadrivalent (Influenza Vaccine) in Pregnant Women and Their Offspring
Brief Title: Surveillance Study to Assess the Safety of Flublok Quadrivalent (Influenza Vaccine) in Pregnant Women and Their Offspring
Acronym: VAP00007
Status: Completed | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: VAP00007
Record Dates: First submitted 2020-07-02; First posted 2020-07-08 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 1: Pregnant women from the VAP00003 Study and their offspring - Pregnant women from the VAP00003 Study (NCT03694392) between September 2018 and May 2020 (2 influenza seasons), and infants born from this cohort of pregnant women
  Interventions: Biological: Flublok Quadrivalent influenza vaccine RIV4; Biological: Standard-dose quadrivalent inactivated influenza vaccine SD-IIV4

INTERVENTIONS:
Biological: Flublok Quadrivalent influenza vaccine RIV4 — Route of administration: Intramuscular
  Other Names: RIV4
Biological: Standard-dose quadrivalent inactivated influenza vaccine SD-IIV4 — Route of administration: Intramuscular
  Other Names: SD-IIV4

SUMMARY:
Primary Objective:

To evaluate the safety of Flublok Quadrivalent influenza vaccine in pregnant women included in the VAP00003 Study (NCT03694392) and their offspring exposed during pregnancy or up to 28 days preceding the estimated date of conception with regards to pregnancy, birth, and neonatal/infant outcomes

Secondary Objective:

DETAILED DESCRIPTION:
Data will be recorded prospectively during the safety follow-up for pregnant women until delivery (or pregnancy outcome, whichever is later), and for infants of pregnant women for 1 year after birth.

ELIGIBILITY:
Inclusion criteria

Pregnant women:

* Laboratory or medical professional confirmation of pregnancy
* Exposure to either Flublok Quadrivalent influenza vaccine or standard-dose quadrivalent inactivated influenza vaccine (SD-IIV4) in the VAP00003 Study during pregnancy or within 28 days preceding conception

Offspring:

* Infants delivered by pregnant women who satisfy the criteria above Exclusion criteria
* Documented receipt of any other influenza vaccine at any other time during the pregnancy

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Max Age: 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women were not randomized. A modified-cluster randomization scheme was used. Facilities were assigned to blocks and were randomized within blocks, ensuring that roughly half the facilities within each block initially administer one vaccine of the 2 vaccines planned in the study, and the other half administer the alternate vaccine. Iteratively, over time, the vaccine administered within each facility will then alternate.
Sampling Method: Probability Sample
Enrollment: 96175 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Incidence Rates of Pregnancy Outcome Events | From start of pregnancy or up to 28 days prior to conception until delivery or pregnancy outcome
  Pregnancy outcome events: spontaneous abortion, preterm labor, stillbirth/Fetal death, congenital/fetal anomalies detected during pregnancy, eclampsia, and placental abruption
Incidence Rates of Birth Events | At birth
  Preterm birth, low birth weight or small for gestational age observed or diagnosed at birth
Incidence Rates of Neonatal/ Infant Outcomes | From birth to Day 365 post-birth
  Neonatal/ infant outcomes: infant death, any congenital anomalies detected after delivery, and failure to thrive

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (1):
- Kaiser Permanente Northern California, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org